CLINICAL TRIAL: NCT00568906
Title: Microarray Analysis of Gene Expression and Identification of Progenitor Cells in Lung Carcinoma
Status: Terminated | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: LUN0011; 76094 (Other: Stanford University Alternate IRB Approval Number); SU-11062007-807 (Other: Stanford University); 12472 (Other: Stanford IRB)
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Carcinoma, Giant Cell; Carcinoma, Non-Small-Cell Lung; Lung Cancer
MeSH Terms: conditions — Carcinoma, Giant Cell; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Lung tissue or pleural fluid.

SUMMARY:
This study will help us understand the gene expression profiles of lung cancer. We will identify genes related to lung cancer development, their growth and metastasis to the lung. In addition, we will examine the role nicotine in the development and progression of lung tumors of smokers, ex-smokers, non-smokers on supplemental nicotine and non smokers with no exposure to nicotine.

ELIGIBILITY:
Inclusion Criteria:Adults with non small cell lung cancer Exclusion Criteria:NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who agree to participate in this study will be those who are undergoing wedge resection, lobectomy on pneumonectomy for clinically diagnosed lung carcinoma or metastatic tumors to the lung, or who are undergoing therapeutic or diagnostic thoracentesis for malignant pleural effusion.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2002-02; Primary Completion 2010-11-30 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
identify genes related to lung cancer development, their growth and metastasis to the lung. | day one

CONTACTS AND LOCATIONS:
Overall Officials: Daya Upadhyay, Principal Investigator — Stanford University; Glenn D. Rosen, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States